CLINICAL TRIAL: NCT04524130
Title: The Effect of Intraoperative Lidocaine Infusion and Intraoperative Lidocaine Combined With Ketamine Infusion on Opioid Consumption After Laparoscopic Bariatric Surgery: A Randomized Controlled Trial
Brief Title: Intraoperative Lidocaine and Combined With Ketamine on Opioid After Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 610/2563(IRB3)
Record Dates: First submitted 2020-07-29; First posted 2020-08-24 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Laparoscopic Bariatric Surgery
MeSH Terms: interventions — Lidocaine; Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lidocaine and Ketamine (Experimental): Participants in this arm will receive intra-operative lidocaine and ketamine infusion as adjunctive drugs for pain control. All medication is dosed based on calculated lean body weight (LBW) by Janmahasatian formula.
  Interventions: Drug: Lidocaine Hydrochloride; Drug: Ketamine
- Lidocaine (Active Comparator): Participants in this arm will receive only intra-operative ketamine infusion as adjunctive drugs for pain control. All medication is dosed based on calculated lean body weight (LBW) by Janmahasatian formula.
  Interventions: Drug: Lidocaine Hydrochloride; Drug: Placebo
- Placebo (Placebo Comparator): Participants in this arm will receive normal saline, same volume as lidocaine and ketamine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — lidocaine will be given 1.5 mg/kg bolus at induction then 2mg/kg/hr until the end of surgery.
  Other Names: Li
  Arms: Lidocaine; Lidocaine and Ketamine
Drug: Ketamine — Ketamine will be given 0.35 mg/kg bolus at induction then 0.2 mg/kg/hr until the end of surgery.
  Other Names: Ke
  Arms: Lidocaine and Ketamine
Drug: Placebo — Normal saline will be given with the same rate of lidocaine or ketamine.
  Other Names: Normal Saline
  Arms: Lidocaine; Placebo

SUMMARY:
The most effective long-term treatment for obesity is bariatric surgery, however, postoperative pain control is challenging in these group of population. Opioid-sparing technique with multimodal analgesia is recommended but the evidence supported is still limited. Multimodal analgesia, particularly lidocaine and ketamine, has been used effectively in various type of surgery. However, the evidence supported their use in obese patients undergoing bariatric surgery is limited.

DETAILED DESCRIPTION:
The prevalence of obesity and associated diseases have been increasing in recent decades. From 1980 to 2013, the number of adults with BMI more than 25 kg/m2 increased from 28.8% to 36.9% in men, and from 29.8% to 38% in women. According to World Health Organization (WHO), the prevalence of overweight among adults in Thailand in 2016 was 32.6%, markedly increased from 2011 which was 23.9%. To date, the most effective long-term treatment for obesity is bariatric surgery because of significantly reducing body fat, the development of new obesity-related conditions, and overall mortality. However, postoperative complications, particularly respiratory complication, are concerned because obesity is associated with respiratory compromise and sleep-disordered breathing. The 2016 guideline for perioperative care in bariatric surgery developed by enhanced recovery after surgery (ERAS) society state that, regarding to current evidence, there is no specific anesthetic agents or techniques for bariatric surgery, however, multimodal analgesia should be used to reduce opioid consumption and opioid-related complications such as respiratory depression, postoperative nausea and vomiting and ileus. Moreover, several studies supported opioid-sparing technique to avoid respiratory complications.

Intravenous lidocaine is widely used to reduce postoperative pain and to reduce perioperative opioid as a multimodal analgesia. From Cochrane review, perioperative lidocaine can decrease pain at rest, postoperative ileus and postoperative nausea and vomiting in elective and urgent surgery. Few trials in obese patients underwent laparoscopic bariatric surgery found that lidocaine infusion can decrease opioid consumption. However, the supported evidence is still limit. Ketamine has been used for postoperative analgesia as well, as an effective adjunct to decrease opioid consumption in various types of surgery, including open bariatric surgery. Moreover, the recent retrospective study (Tovikkai P, in press) found that there was a positive interaction between intraoperative lidocaine infusion and ketamine for decreasing opioid consumption in obese patients underwent laparoscopic bariatric surgery. However, the benefit of lidocaine and ketamine for postoperative pain in obese patients underwent laparoscopic bariatric surgery is still debated.

Therefore, we designed this study to examine the effect of intraoperative lidocaine infusion and intraoperative lidocaine infusion combined with intraoperative low-dose ketamine infusion on opioid consumption in obese patients undergoing laparoscopic bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults patients age older than 18 years.
2. Body mass index more than 30 kg/m2.
3. Scheduled for laparoscopic bariatric surgery, including laparoscopic sleeve gastrectomy, robotic-assisted laparoscopic sleeve gastrectomy, laparoscopic Roux-en-Y gastric bypass surgery or robotic-assisted laparoscopic gastric bypass.

Exclusion Criteria:

1. Patient refusal.
2. Inability to communicate or read in Thai language.
3. Allergic to lidocaine or ketamine.
4. History of opioid use within 2 weeks before surgery
5. Cardiovascular disorder, including high grade atrioventricular block (second degree or third degree), history of coronary artery disease, poor controlled hypertension.
6. History of stroke, intracranial hemorrhage or intracranial mass
7. Cognitive impairment
8. Schizophrenia or history of antipsychotic drugs
9. Pregnant or breast-feeding patients
10. Conversion to open surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 24-hour
  Opioid consumption at 24 hr post-operation using Morphine Milligram equivalents(MME)
Score of post-extubation cough | up to 24 hours (at extubation period after surgery finished)
  post-extubation cough graded by care giver using modified Minogue scales, which defined grade1 as no coughing or muscular stiffness, grade 2 as coughing once or twice, or transient cough response to removal of tracheal tube that resolved with extubation, grade 3 as ≤ 3 coughs lasting 1-2 seconds, or total duration of coughing last ≤ 5 seconds and grade 4 as ≥ 4 coughs with each lasting > 2 seconds, total duration of coughing last > 5 seconds.

SECONDARY OUTCOMES:
operative time | intraoperative (since the incision started until finished the last suture)
  time since incision started until the last suture done recorded in minutes.
anesthetic time | intraoperative (since anesthetic started until patient out of the operating room)
  time since anesthetic started until finished and patient out of room recorded in minutes.
the length of hospital stay | until 30-day postoperation
  time since admission until discharge recorded in hours.
numbers of participants with postoperative complications | until 30-day postoperation
  cardiac arrhythmia, myocardial infarction, respiratory compromised, reintubation, readmission.
Score of sore throat | assess at 24-hour post-operation
  sore throat score grading by self-assessment score, which defined grade 0 as no sore throat, grade 1 as minimal sore throat, grade 2 as moderate sore throat and grade 3 as severe sore throat.

CONTACTS AND LOCATIONS:
Overall Officials: Parichat Tovikkai, Principal Investigator — Mahidol University
Locations (1):
- Faculty of medicine Siriraj hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830
- [Background] Jitnarin N, Kosulwat V, Rojroongwasinkul N, Boonpraderm A, Haddock CK, Poston WS. Prevalence of overweight and obesity in Thai population: results of the National Thai Food Consumption Survey. Eat Weight Disord. 2011 Dec;16(4):e242-9. doi: 10.1007/BF03327467. PMID 22526130
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Lukosiute A, Karmali A, Cousins JM. Anaesthetic Preparation of Obese Patients: Current Status on Optimal Work-up. Curr Obes Rep. 2017 Sep;6(3):229-237. doi: 10.1007/s13679-017-0268-5. PMID 28707209
- [Background] Ortiz VE, Kwo J. Obesity: physiologic changes and implications for preoperative management. BMC Anesthesiol. 2015 Jul 4;15:97. doi: 10.1186/s12871-015-0079-8. PMID 26141622
- [Background] Thorell A, MacCormick AD, Awad S, Reynolds N, Roulin D, Demartines N, Vignaud M, Alvarez A, Singh PM, Lobo DN. Guidelines for Perioperative Care in Bariatric Surgery: Enhanced Recovery After Surgery (ERAS) Society Recommendations. World J Surg. 2016 Sep;40(9):2065-83. doi: 10.1007/s00268-016-3492-3. PMID 26943657
- [Background] King AB, Spann MD, Jablonski P, Wanderer JP, Sandberg WS, McEvoy MD. An enhanced recovery program for bariatric surgical patients significantly reduces perioperative opioid consumption and postoperative nausea. Surg Obes Relat Dis. 2018 Jun;14(6):849-856. doi: 10.1016/j.soard.2018.02.010. Epub 2018 Feb 13. PMID 29555468
- [Background] Feld JM, Laurito CE, Beckerman M, Vincent J, Hoffman WE. Non-opioid analgesia improves pain relief and decreases sedation after gastric bypass surgery. Can J Anaesth. 2003 Apr;50(4):336-41. doi: 10.1007/BF03021029. English, French. PMID 12670809
- [Background] Soto G, Naranjo Gonzalez M, Calero F. Intravenous lidocaine infusion. Rev Esp Anestesiol Reanim (Engl Ed). 2018 May;65(5):269-274. doi: 10.1016/j.redar.2018.01.004. Epub 2018 Feb 26. English, Spanish. PMID 29496229
- [Background] Weibel S, Jelting Y, Pace NL, Helf A, Eberhart LH, Hahnenkamp K, Hollmann MW, Poepping DM, Schnabel A, Kranke P. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery in adults. Cochrane Database Syst Rev. 2018 Jun 4;6(6):CD009642. doi: 10.1002/14651858.CD009642.pub3. PMID 29864216
- [Background] De Oliveira GS Jr, Duncan K, Fitzgerald P, Nader A, Gould RW, McCarthy RJ. Systemic lidocaine to improve quality of recovery after laparoscopic bariatric surgery: a randomized double-blinded placebo-controlled trial. Obes Surg. 2014 Feb;24(2):212-8. doi: 10.1007/s11695-013-1077-x. PMID 24036842
- [Background] Sakata RK, de Lima RC, Valadao JA, Leal PC, Moura EC, Cruz VP, de Oliveira CM. Randomized, Double-Blind Study of the Effect of Intraoperative Intravenous Lidocaine on the Opioid Consumption and Criteria for Hospital Discharge After Bariatric Surgery. Obes Surg. 2020 Apr;30(4):1189-1193. doi: 10.1007/s11695-019-04340-2. PMID 31858394
- [Background] Gupta C, Valecha UK, Singh SP, Varshney M. Systemic lidocaine versus ultrasound-guided transversus abdominis plane block for postoperative analgesia: A comparative randomised study in bariatric surgical patients. Indian J Anaesth. 2020 Jan;64(1):31-36. doi: 10.4103/ija.IJA_430_19. Epub 2020 Jan 7. PMID 32001906
- [Background] Laskowski K, Stirling A, McKay WP, Lim HJ. A systematic review of intravenous ketamine for postoperative analgesia. Can J Anaesth. 2011 Oct;58(10):911-23. doi: 10.1007/s12630-011-9560-0. Epub 2011 Jul 20. PMID 21773855
- [Background] Radvansky BM, Shah K, Parikh A, Sifonios AN, Le V, Eloy JD. Role of ketamine in acute postoperative pain management: a narrative review. Biomed Res Int. 2015;2015:749837. doi: 10.1155/2015/749837. Epub 2015 Oct 1. PMID 26495312
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Sollazzi L, Modesti C, Vitale F, Sacco T, Ciocchetti P, Idra AS, Tacchino RM, Perilli V. Preinductive use of clonidine and ketamine improves recovery and reduces postoperative pain after bariatric surgery. Surg Obes Relat Dis. 2009 Jan-Feb;5(1):67-71. doi: 10.1016/j.soard.2008.09.018. Epub 2008 Oct 17. PMID 19095506
- [Background] Tovikkai P, Rogers SJ, Cello JP, Mckay RE. Intraoperative lidocaine infusion and 24-hour postoperative opioid consumption in obese patients undergoing laparoscopic bariatric surgery. Surg Obes Relat Dis. 2020 Aug;16(8):1124-1132. doi: 10.1016/j.soard.2020.04.026. Epub 2020 May 4. PMID 32553616
- [Background] Wang J, Echevarria GC, Doan L, Ekasumara N, Calvino S, Chae F, Martinez E, Robinson E, Cuff G, Franco L, Muntyan I, Kurian M, Schwack BF, Bedrosian AS, Fielding GA, Ren-Fielding CJ. Effects of a single subanaesthetic dose of ketamine on pain and mood after laparoscopic bariatric surgery: A randomised double-blind placebo controlled study. Eur J Anaesthesiol. 2019 Jan;36(1):16-24. doi: 10.1097/EJA.0000000000000860. PMID 30095550